CLINICAL TRIAL: NCT06717672
Title: Efficacy of Lidocaine in Decreasing Perioperative Analgesic Opioids Requirement After Ambulatory Surgery
Brief Title: Effect of Lidocaine in Reducing Opioids Requirement in Day Care Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Liaquat National Hospital & Medical College (Other)
Responsible Party: Principal Investigator, Hanesh Tanwani, Principal Investigator, Liaquat National Hospital & Medical College
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ANS-2021-192-2750
Record Dates: First submitted 2024-11-30; First posted 2024-12-05 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Pain; Post-operative Pain Control; Post-operative Pain
Keywords: Lidocaine; Opiods; Peri-operative pain; Decrease Opioid requirement; Ambulatory surgeries
MeSH Terms: conditions — Pain; Pain, Postoperative | interventions — Lidocaine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Active Comparator): intervention group recieve inj lidocaine
  Interventions: Drug: Lidocaine 2% without vessel constrictor
- Control group (Placebo Comparator): control group receive Normal saline
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Lidocaine 2% without vessel constrictor — 1. _Lidocaine 2% provides rapid and effective local anesthesia for minor surgical procedures, such as biopsies, excisions, and suturing.
  2. _Pain relief_: Lidocaine 2% has been shown to provide significant pain relief in patients with acute pain, such as post-operative pain, trauma, and burns.
  3. _Reducing pain intensity_: Lidocaine 2% has been shown to reduce pain intensity by 30-50% in various clinical studies.
  Arms: Intervention group
Drug: Normal Saline — Normal saline used is an iv fluid given for fluid replacement
  Arms: Control group

SUMMARY:
1. *Reduced opioid consumption
2. *Decreased pain scores
3. *Fewer opioid-related side effects
4. *Improved patient satisfaction

DETAILED DESCRIPTION:
Studies have shown that lidocaine can reduce opioid consumption by 20-50% in the perioperative period.

Studies have shown that lidocaine can reduce opioid consumption by 20-50% in the perioperative period.

By reducing opioid consumption, lidocaine can also decrease the incidence of opioid-related side effects, such as nausea, vomiting, and respiratory depression.

Lidocaine's analgesic effects can improve patient satisfaction and reduce anxiety related to pain

ELIGIBILITY:
Inclusion Criteria:

* ASA 1 and 2
* patient age between 18 and 65 years
* Patient undergoing ambulatory surgeries

Exclusion Criteria:

* Pregnant women
* Allergic to Lidocaine Patient who had fever and treated with antibiotic and steroid in last month

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2023-11-05 (Actual); Primary Completion 2024-05-10 (Actual); Study Completion 2024-05-10 (Actual)

PRIMARY OUTCOMES:
Peri-operative pain | at 2 hours, 4 hours, 6 hours
  Visual Analog pain scale to rate pain scale comprises 0 to 10 score 0 minimum to 10 Maximum

CONTACTS AND LOCATIONS:
Overall Officials: Hanesh Tanwani Dr Hanesh Tanwani, Principal Investigator — Liaquat National Hospital and Medical College
Locations (1):
- Liaquat National Hospital and Medical College, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No
*Informed consent*: Participants may not have provided informed consent for their data to be shared, which could raise ethical concerns.
  Patient confidentiality*: Sharing IPD could compromise patient confidentiality and anonymity, potentially harming participants or their families.

REFERENCES:
- See also: Systemic lidocaine decreased the perioperative opioid analgesic requirements but failed to reduce discharge time after ambulatory surgery Allannah McKay 1, Antje Gottschalk, Annette Ploppa, Marcel E Durieux, Danja S Groves — https://pubmed.ncbi.nlm.nih.gov/19923506/